CLINICAL TRIAL: NCT02648347
Title: Phase 3, Randomized, Open-Label, Active-Controlled Study Evaluating the Efficacy and Safety of Oral Vadadustat for the Correction of Anemia in Subjects With Non-Dialysis-Dependent Chronic Kidney Disease (NDD-CKD) (PRO2TECT-CORRECTION)
Brief Title: Study to Evaluate Vadadustat for the Correction of Anemia in Participants With Non-dialysis-dependent Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0014; 2015-004265-81 (EudraCT Number)
Record Dates: First submitted 2016-01-04; First posted 2016-01-07 (Estimated); Results first posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Anemia; Non-Dialysis-Dependent Chronic Kidney Disease
Keywords: Vadadustat; AKB-6548; Chronic kidney disease; anemia; CKD; chronic renal insufficiency; renal impairment; erythropoietin; kidney; renal; oral anemia treatment; hemoglobin; hypoxia-inducible factor; HIF; hypoxia-inducible factor prolyl-hydroxylase inhibitor; HIF-PHI; efficacy; safety; Phase 3; cardiovascular; NDD-CKD
MeSH Terms: conditions — Anemia; Renal Insufficiency, Chronic; Renal Insufficiency | interventions — vadadustat; Darbepoetin alfa

STUDY DESIGN:
Masking Description: Sponsor was blinded during the study
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vadadustat (Experimental)
  Interventions: Drug: Vadadustat
- Darbepoetin alfa (Active Comparator)
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Vadadustat — Oral dose administered once daily for ≥36 weeks. Dose adjustment based on hemoglobin level as defined in the protocol.
  Other Names: AKB-6548
  Arms: Vadadustat
Drug: Darbepoetin alfa — Subcutaneous or intravenous dose administered for ≥36 weeks. Initial dose based on the current package insert for investigational sites in the United States (US), and the Summary of Product Characteristics for all other investigational sites (non-US) for adult participants with chronic kidney disease not on dialysis.
  Other Names: Aranesp
  Arms: Darbepoetin alfa

SUMMARY:
A multicenter, randomized, open-label, active-controlled Phase 3 study for the correction of anemia and maintenance of hemoglobin (Hb) in participants with Non-Dialysis-Dependent Chronic Kidney Disease (NDD-CKD)

DETAILED DESCRIPTION:
This is a multicenter, randomized, open-label, active-controlled Phase 3 study of the efficacy and safety of vadadustat versus Darbepoetin alfa for the correction of anemia and maintenance of Hb in participants with NDD-CKD

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Diagnosis of chronic kidney disease (CKD) with an estimated glomerular filtration rate ≤60 milliliters per minute per 1.73 square meter (mL/min/1.73 m^2) at Screening and not expected to start dialysis within 6 months of Screening
* Mean Screening hemoglobin <10.0 grams per deciliter (g/dL)
* Serum ferritin ≥100 nanograms per milliliter (ng/mL) and transferrin saturation (TSAT) ≥20% during Screening

Exclusion Criteria:

* Anemia due to a cause other than CKD or participants with active bleeding or recent blood loss
* Red blood cell transfusion within 8 weeks prior to randomization.
* Any erythropoietic stimulating agent within 8 weeks prior to randomization
* Uncontrolled hypertension
* Severe heart failure at Screening (New York Heart Association Class IV)
* Acute coronary syndrome (hospitalization for unstable angina or myocardial infarction), surgical or percutaneous intervention for coronary, cerebrovascular, or peripheral artery disease (aortic or lower extremity), surgical or percutaneous valvular replacement or repair, sustained ventricular tachycardia, hospitalization for heart failure, or stroke within 12 weeks prior to or during Screening
* Hypersensitivity to Darbepoetin or Vadadustat or to any of their excipients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1751 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2020-06-04 (Actual); Study Completion 2020-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chief Medical Officer, Study Director — Akebia Therapeutics Inc.
Locations (355):
- United States (176):
  - Research Site, Huntsville, Alabama
  - Research Site, Tuscumbia, Alabama
  - Research Site, Glendale, Arizona
  - Research Site, Mesa, Arizona
  - Research Site, Phoenix, Arizona
  - Research Site, Tucson, Arizona
  - Research Site, Anaheim, California
  - Research Site, Bakersfield, California
  - Research Site #1, Chula Vista, California
  - Research Site #2, Chula Vista, California
  - Research Site #1, Fountain Valley, California
  - Research Site #2, Fountain Valley, California
  - Research Site, Glendale, California
  - Research Site, Granada Hills, California
  - Research Site, La Mesa, California
  - Research Site, Laguna Hills, California
  - Research Site, Long Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Lynwood, California
  - Research Site #2, Northridge, California
  - Research Site, Northridge, California
  - Research Site, Riverside, California
  - Research Site, Roseville, California
  - Research Site, Sacramento, California
  - Research Site, Salinas, California
  - Research Site, San Diego, California
  - Research Site #1, San Dimas, California
  - Research Site #2, San Dimas, California
  - Research Site, Santa Ana, California
  - Research Site, Santa Monica, California
  - Research Site, Sherman Oaks, California
  - Research Site, Thousand Oaks, California
  - Research Site, Upland, California
  - Research Site #1, Whittier, California
  - Research Site #2, Whittier, California
  - Research Site, Arvada, Colorado
  - Research Site, Denver, Colorado
  - Research Site, Westminster, Colorado
  - Research Site, New Haven, Connecticut
  - Research Site, Stamford, Connecticut
  - Research Site, Waterbury, Connecticut
  - Research Site, Bradenton, Florida
  - Research Site, Brandon, Florida
  - Research Site, Cooper City, Florida
  - Research Site #1, Coral Gables, Florida
  - Research Site #2, Coral Gables, Florida
  - Research Site, Coral Springs, Florida
  - Research Site, Doral, Florida
  - Research Site, Fort Myers, Florida
  - Research Site, Hialeah, Florida
  - Research Site #1, Hialeah, Florida
  - Research Site #2, Hialeah, Florida
  - Research Site #3, Hialeah, Florida
  - Research Site #1, Hollywood, Florida
  - Research Site #2, Hollywood, Florida
  - Research Site, Jacksonville, Florida
  - Research Site #1, Jacksonville, Florida
  - Research Site #2, Jacksonville, Florida
  - Research Site, Lake Worth, Florida
  - Research Site, Lauderdale Lakes, Florida
  - Research Site, Miami, Florida
  - Research Site #1, Miami, Florida
  - Research Site #2, Miami, Florida
  - Research Site, Miami Beach, Florida
  - Research Site, Miami Lakes, Florida
  - Research Site, Miami Springs, Florida
  - Research Site, Pembroke Pines, Florida
  - Research Site, Pompano Beach, Florida
  - Research Site, Sweetwater, Florida
  - Research Site, Tampa, Florida
  - Research Site, Atlanta, Georgia
  - Research Site #1, Augusta, Georgia
  - Research Site #2, Augusta, Georgia
  - Research Site, Columbus, Georgia
  - Research Site #1, Columbus, Georgia
  - Research Site #2, Columbus, Georgia
  - Research Site #1, Lawrenceville, Georgia
  - Research Site #2, Lawrenceville, Georgia
  - Research Site, Macon, Georgia
  - Research Site, Meridian, Idaho
  - Research Site, Chicago, Illinois
  - Research Site, Evanston, Illinois
  - Research Site, McHenry, Illinois
  - Research Site, Peoria, Illinois
  - Research Site, Anderson, Indiana
  - Research Site, Fort Wayne, Indiana
  - Research Site, Jeffersonville, Indiana
  - Research Site #1, Merrillville, Indiana
  - Research Site #2, Merrillville, Indiana
  - Research Site, Michigan City, Indiana
  - Research Site, Monroe, Louisiana
  - Research Site, New Orleans, Louisiana
  - Research Site #1, Shreveport, Louisiana
  - Research Site, Shreveport, Louisiana
  - Research Site, Portland, Maine
  - Research Site, Baltimore, Maryland
  - Research Site, Greenbelt, Maryland
  - Research Site, Takoma Park, Maryland
  - Research Site, Methuen, Massachusetts
  - Research Site, Plymouth, Massachusetts
  - Research Site, Detroit, Michigan
  - Research Site, Pontiac, Michigan
  - Research Site, Roseville, Michigan
  - Research Site, Saint Paul, Minnesota
  - Research Site, Gulfport, Mississippi
  - Research Site, Columbia, Missouri
  - Research Site, Kansas City, Missouri
  - Research Site, St Louis, Missouri
  - Research Site, Butte, Montana
  - Research Site, Lincoln, Nebraska
  - Research Site, Omaha, Nebraska
  - Research Site #1, Las Vegas, Nevada
  - Research Site #2, Las Vegas, Nevada
  - Research Site, Portsmouth, New Hampshire
  - Research Site, Berlin, New Jersey
  - Research Site, Voorhees Township, New Jersey
  - Research Site, Albuquerque, New Mexico
  - Research Site, Santa Fe, New Mexico
  - Research Site, Flushing, New York
  - Research Site, Laurelton, New York
  - Research Site, New York, New York
  - Research Site, The Bronx, New York
  - Research Site, Asheville, North Carolina
  - Research Site #1, Greenville, North Carolina
  - Research Site #2, Greenville, North Carolina
  - Research Site, Kinston, North Carolina
  - Research Site, Morehead City, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Akron, Ohio
  - Research Site, Cincinnati, Ohio
  - Research Site, Dayton, Ohio
  - Research Site, Marion, Ohio
  - Research Site, Maumee, Ohio
  - Research Site, Portland, Oregon
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, East Providence, Rhode Island
  - Research Site, Anderson, South Carolina
  - Research Site, Orangeburg, South Carolina
  - Research Site, West Columbia, South Carolina
  - Research Site, Chattanooga, Tennessee
  - Research Site, Knoxville, Tennessee
  - Research Site, Memphis, Tennessee
  - Research Site, Nashville, Tennessee
  - Research Site, Arlington, Texas
  - Research Site, Dallas, Texas
  - Research Site, DeSoto, Texas
  - Research Site, El Paso, Texas
  - Research Site, Fort Worth, Texas
  - Research Site, Gonzales, Texas
  - Research Site, Greenville, Texas
  - Research Site #1, Houston, Texas
  - Research Site #2, Houston, Texas
  - Research Site, Houston, Texas
  - Research Site, Lewisville, Texas
  - Research Site #1, McAllen, Texas
  - Research Site #2, McAllen, Texas
  - Research Site, McKinney, Texas
  - Research Site, Plano, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sherman, Texas
  - Research Site, Victoria, Texas
  - Research Site, Clinton, Utah
  - Research Site, Salt Lake City, Utah
  - Research Site, Alexandria, Virginia
  - Research Site, Arlington, Virginia
  - Research Site, Danville, Virginia
  - Research Site, Hampton, Virginia
  - Research Site, Lansdowne Town Center, Virginia
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia
  - Research Site, Salem, Virginia
  - Research Site, Woodbridge, Virginia
  - Research Site, Tacoma, Washington
  - Research Site, Wenatchee, Washington
  - Research Site, Madison, Wisconsin
- Argentina (17):
  - Research Site, Bahía Blanca, Buenos Aires
  - Research Site, Junín, Buenos Aires
  - Research Site, Mar del Plata, Buenos Aires
  - Research Site, Pergamino, Buenos Aires
  - Research Site, Ramos Mejía, Buenos Aires
  - Research Site, San Miguel, Buenos Aires
  - Research Site, San Nicolás de los Arroyos, Buenos Aires
  - Research Site, Sarandí, Buenos Aires
  - Research Site, Temperley, Buenos Aires
  - Research Site, Godoy Cruz, Mendoza Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
  - Research Site, Ciudad Autonoma Buenos Aires
  - Research Site, Corrientes
  - Research Site, Córdoba
  - Research Site, Salta
  - Research Site, San Luis
- Australia (10):
  - Research Site, Camperdown, New South Wales
  - Research Site, Liverpool, New South Wales
  - Research Site, Cairns, Queensland
  - Research Site, Gold Coast, Queensland
  - Research Site, Herston, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Bedford Park, South Australia
  - Research Site, Box Hill, Victoria
  - Research Site, Nedlands, Western Australia
  - Research Site, Perth, Western Australia
- Brazil (22):
  - Research Site, Fortaleza, Ceará
  - Research Site, Vitória, Espírito Santo
  - Research Site, Feira de Santana, Estado de Bahia
  - Research Site, Itabuna, Estado de Bahia
  - Research Site, Belo Horizonte, Minas Gerais
  - Research Site, Juiz de Fora, Minas Gerais
  - Research Site, Curitiba, Paraná
  - Research Site #1, Curitiba, Paraná
  - Research Site #2, Curitiba, Paraná
  - Research Site, Maringá, Paraná
  - Research Site, Rio de Janeiro, Rio Do Janeiro
  - Research Site, Canoas, Rio Grande do Sul
  - Research Site, Caxias do Sul, Rio Grande do Sul
  - Research Site, Passo Fundo, Rio Grande do Sul
  - Research Site, Porto Alegre, Rio Grande do Sul
  - Research Site, Criciúma, Santa Catarina
  - Research Site, Joinville, Santa Catarina
  - Research Site, Botucatu, São Paulo
  - Research Site, Campinas, São Paulo
  - Research Site, Santo André, São Paulo
  - Research Site, São Bernardo do Campo, São Paulo
  - Research Site, São Paulo, São Paulo
- Bulgaria (13):
  - Research Site, Dobrich
  - Research Site, Lom
  - Research Site, Silistra
  - Research Site, Sliven
  - Research Site, Smolyan
  - Research Site, Sofia
  - Research Site #1, Sofia
  - Research Site #2, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
  - Research Site #1, Veliko Tarnovo
  - Research Site #2, Veliko Tarnovo
  - Research Site, Vidin
- Research Site, Pontoise, Val d'Oise, France
- Hungary (14):
  - Research Site #1, Baja
  - Research Site #2, Baja
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Debrecen
  - Research Site, Hódmezővásárhely
  - Research Site, Kalocsa
  - Research Site, Kaposvár
  - Research Site, Kecskemét
  - Research Site, Kistarcsa
  - Research Site, Nyíregyháza
  - Research Site, Pécs
  - Research Site, Szeged
  - Research Site, Szigetvár
- Israel (5):
  - Research Site, Ashkelon
  - Research Site, Haifa
  - Research Site, Nahariya
  - Research Site, Ramat Gan
  - Research Site, Rishon LeZiyyon
- Italy (13):
  - Research Site, Piedimonte Matese, Caserta
  - Research Site, San Giovanni Rotondo, Foggia
  - Research Site, Bari
  - Research Site, Bergamo
  - Research Site, Cremona
  - Research Site, Genova
  - Research Site, Lecco
  - Research Site, Milan
  - Research Site, Napoli
  - Research Site, Parma
  - Research Site, Pavia
  - Research Site, Roma
  - Research Site, Siena
- Malaysia (2):
  - Research Site, Kota Bharu, Kelantan
  - Research Site, Kuantan, Pahang
- Mexico (13):
  - Research Site, Acapulco de Juárez, Guerrero
  - Research Site, Pachuca, Hidalgo
  - Research Site, Guadalajara, Jalisco
  - Research Site, Zapopan, Jalisco
  - Research Site, Mexico City, Mexico City
  - Research Site, Morelia, Michoacán
  - Research Site, Monterrey, Nuevo León
  - Research Site, San Juan del Río, Querétaro
  - Research Site, Culiacán, Sinaloa
  - Research Site, Mazatlán, Sinaloa
  - Research Site, Chihuahua City
  - Research Site, Durango
  - Research Site, Veracruz
- New Zealand (2):
  - Research Site, Hamilton
  - Research Site, New Plymouth
- Poland (4):
  - Research Site, Lodz
  - Research Site, Nowa Sól
  - Research Site, Warsaw
  - Research Site, Wroclaw
- Research Site, Caguas, Puerto Rico
- Russia (12):
  - Research Site, Kazan'
  - Research Site, Kemerovo
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Petrozavodsk
  - Research Site, Pushkin
  - Research Site, Saint Petersburg
  - Research Site, Tomsk
  - Research Site, Tosno
  - Research Site, Yaroslavl
- South Africa (15):
  - Research Site, Port Elizabeth, Eastern Cape
  - Research Site, Bloemfontein, Free State
  - Research Site, Winnie Mandela, Free State
  - Research Site #1, Pretoria, Gauteng
  - Research Site #2, Pretoria, Gauteng
  - Research Site, Pretoria, Gauteng
  - Research Site, Vereeniging, Gauteng
  - Research Site #1, Durban, KwaZulu-Natal
  - Research Site #2, Durban, KwaZulu-Natal
  - Research Site, Durban, KwaZulu-Natal
  - Research Site, Tongaat, KwaZulu-Natal
  - Research Site, Cape Town, Western Cape
  - Research Site, George, Western Cape
  - Research Site, Somerset West, Western Cape
  - Research Site, Worcester, Western Cape
- South Korea (5):
  - Research Site, Bucheon-si, Gyeonggi-do
  - Research Site, Guri-si, Gyeonggi-do
  - Research Site, Busan
  - Research Site, Daegu
  - Research Site, Seoul
- Spain (11):
  - Research Site, Elche, Alicante
  - Research Site, Torrevieja, Alicante
  - Research Site, Palma de Mallorca, Balearic Islands
  - Research Site, L'Hospitalet de Llobregat, Barcelona
  - Research Site, Málaga, Málaga
  - Research Site, Almería
  - Research Site, Badajoz
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
- Ukraine (11):
  - Research Site, Dnipro
  - Research Site, Ivano-Frankivsk
  - Research Site, Kharkiv
  - Research Site, Kropyvnytskyi
  - Research Site, Kyiv
  - Research Site, Lviv
  - Research Site, Mykolaiv
  - Research Site, Odesa
  - Research Site, Vinnytsia
  - Research Site, Zaporizhzhia
  - Research Site, Zhytomyr
- United Kingdom (8):
  - Research Site, Aberdeen, Grampian Region
  - Research Site, London, Greater London
  - Research Site, Salford, Greater Manchester
  - Research Site, Stevenage, Hertfordshire
  - Research Site, Leicester, Leicestershire
  - Research Site, Doncaster, South Yorkshire
  - Research Site, Sheffield, South Yorkshire
  - Research Site, Swansea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chertow GM, Eckardt KU, Sarnak MJ, Winkelmayer WC, Agarwal R, Minga T, Luo W, Burke SK. Safety and Efficacy of Vadadustat for the Treatment of CKD-Related Anemia within and outside the United States. J Am Soc Nephrol. 2025 Oct 1;36(10):1984-1997. doi: 10.1681/ASN.0000000708. Epub 2025 May 13. PMID 40359056
- [Derived] Natale P, Palmer SC, Jaure A, Hodson EM, Ruospo M, Cooper TE, Hahn D, Saglimbene VM, Craig JC, Strippoli GF. Hypoxia-inducible factor stabilisers for the anaemia of chronic kidney disease. Cochrane Database Syst Rev. 2022 Aug 25;8(8):CD013751. doi: 10.1002/14651858.CD013751.pub2. PMID 36005278
- [Derived] Chertow GM, Pergola PE, Farag YMK, Agarwal R, Arnold S, Bako G, Block GA, Burke S, Castillo FP, Jardine AG, Khawaja Z, Koury MJ, Lewis EF, Lin T, Luo W, Maroni BJ, Matsushita K, McCullough PA, Parfrey PS, Roy-Chaudhury P, Sarnak MJ, Sharma A, Spinowitz B, Tseng C, Tumlin J, Vargo DL, Walters KA, Winkelmayer WC, Wittes J, Eckardt KU; PRO2TECT Study Group. Vadadustat in Patients with Anemia and Non-Dialysis-Dependent CKD. N Engl J Med. 2021 Apr 29;384(17):1589-1600. doi: 10.1056/NEJMoa2035938. PMID 33913637

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 4708 participants were screened for entry into the study. Of these, 1751 participants were enrolled and randomized into the study.
Groups:
- Vadadustat: Participants were randomized to receive Vadadustat at an initial oral dose of 300 milligrams per day (mg/day). Thereafter, Vadadustat was taken once daily on an outpatient basis. Up-and-down titration to 150, 300, 450, and 600 mg (available tablet strength was administered as the appropriate number of 150 mg tablets) was allowed during the study based on hemoglobin (Hb) level measurements to maintain target Hb levels.
- Darbepoetin Alfa: Participants were randomized to Darbepoetin alfa at an initial dose that was based on the current package insert for investigational sites in the United States (US), and the Summary of Product Characteristics (SmPC) for all other investigational sites (non-US) for adult participants with chronic kidney disease not on dialysis.
Period: Overall Study
Arm/Group | Vadadustat | Darbepoetin Alfa
Started | 879 | 872
Completed | 670 | 675
Not Completed | 209 | 197
Not completed — Death | 174 | 167
Not completed — Withdrawal by Subject | 16 | 9
Not completed — Lost to Follow-up | 18 | 21
Not completed — Missing | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat | Darbepoetin Alfa | Total
Number analyzed (Participants) | 879 | 872 | 1751
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.2 (14.27) | 64.9 (13.71) | 65.0 (13.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 475 | 506 | 981
  Male | 404 | 366 | 770
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 22 | 23 | 45
  Asian | 48 | 37 | 85
  Black or African American | 188 | 172 | 360
  Native Hawaiian or Other Pacific Islander | 6 | 6 | 12
  White | 546 | 571 | 1117
  Not Reported | 5 | 6 | 11
  Reported as Other | 58 | 48 | 106
  Multiple | 6 | 9 | 15
Mean hemoglobin [Mean (Standard Deviation); unit: Grams per deciliter (g/dL)] | 9.113 (0.8015) | 9.142 (0.7790) | 9.128 (0.7903)
Mean estimated glomerular filtration rate [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 21.2 (11.99) | 21.9 (12.60) | 21.5 (12.30)
Number of Participants with History of Diabetes [Count of Participants; unit: Participants] | 507 | 514 | 1021
Number of Participants with NYHA Functional Classification of Heart Failure [Count of Participants; unit: Participants] — The New York Heart Association (NYHA) functional classification serves as a fundamental descriptor of heart failure. NYHA heart failure classes are as follows: Class 0 (no congestive heart failure [CHF]), Class I (No symptoms and no limitation in ordinary physical activity), Class II (Mild symptoms and slight limitation during ordinary activity), Class III (Marked limitation in activity due to symptoms, even during less-than-ordinary activity), and Class IV (Severe limitations. Experiences symptoms even while at rest). NYHA class IV is also an exclusion criteria.
  Participants
    NYHA Class 0 | 613 | 601 | 1214
    NYHA Class I | 136 | 123 | 259
    NYHA Class II | 100 | 119 | 219
    NYHA Class III | 24 | 25 | 49
    NYHA Class IV | 2 | 1 | 3
    NYHA Class Missing | 4 | 3 | 7
Number of Participants with Any History of Heart Failure [Count of Participants; unit: Participants]
  Yes | 36 | 38 | 74
  No | 624 | 609 | 1233
  Missing | 219 | 225 | 444

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hb) to the Average Over the Primary Efficacy Period (Weeks 24 to 36)
Description: The Baseline average was calculated as the average of the Hb values obtained at the screening visit closest to the date of randomization and the randomization visit. The average for the Primary Efficacy Period was calculated as the average Hb value over Weeks 24 to 36. Analysis was conducted using an analysis of covariance (ANCOVA) model with multiple imputation for missing data with Baseline Hb concentration (<9.5 versus ≥9.5 grams per deciliter [g/dL]), geographic region (United States [US] versus European Union [EU] versus Rest of World [ROW]), and New York Heart Association congestive heart failure (NYHA CHF) class (Class 0 [no CHF] or I versus II or III) as covariates.
Time Frame: Baseline; Weeks 24 to 36
Population: Randomized Population: All participants randomized. Analyses of this population were based on the randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 879 | 872
g/dL | 1.43 (0.046) | 1.38 (0.047)
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Treatment comparison: Vadadustat minus Darbepoetin Alfa; Test type: Non-Inferiority — Establishment of non-inferiority was based on a margin of -0.75 g/dL applied to the difference in mean change: Vadadustat minus Darbepoetin alfa; Least squares mean difference = 0.05, 95% CI 2-sided [-0.04 to 0.15], Standard Error of Mean 0.048

2. Primary Outcome: Median Time to First Major Adverse Cardiovascular Event (MACE)
Description: MACE was defined as all-cause mortality, non-fatal myocardial infarction (MI), or non-fatal stroke. The primary safety outcome was positively adjudicated first MACE, which was defined as any death, Endpoint Adjudication Committee (EAC)-confirmed non-fatal MI, or EAC-confirmed non-fatal stroke occurring between the first dose date and each participant's last participation date. PROTECT MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Results and statistical analysis from study AKB-6548-CI-0014 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0014 and AKB-6548-CI-0015 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to Week 208
Population: Safety Population (PRO2TECT): All participants from the PRO2TECT (Non-dialysis-dependent chronic kidney disease [NDD-CKD]) population who received 1 or more doses of study drug. Only those participants with MACE events were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 214 | 192
Weeks | 45.71 [21.71 to 83.14] | 46.71 [25.93 to 85.57]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0014 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per Food and Drug Administration [FDA]) and 1.3 (per European Medicines Agency [EMA]); p = 0.2050, Log Rank; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.955 to 1.412]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Time to first MACE for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 382 and 344 respectively; median time to first event (Q1, Q3) = 50.07 (23.00, 82.86) weeks versus 51.93 (27.79, 91.00) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.0725, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.17, 95% CI 2-sided [1.012 to 1.355]

3. Secondary Outcome: Change From Baseline in Hb to the Average Over the Secondary Efficacy Period (Weeks 40 to 52)
Description: The Baseline average was calculated as the average of the Hb values obtained at the screening visit closest to the date of randomization and the randomization visit. The average for the Secondary Efficacy Period was calculated as the average Hb value over Weeks 40 to 52. Analysis was conducted using an ANCOVA model with multiple imputation for missing data with Baseline Hb concentration (<9.5 versus ≥9.5 g/dL), geographic region (US versus EU versus ROW), and NYHA CHF class (Class 0 [no CHF] or I versus II or III) as covariates.
Time Frame: Baseline; Weeks 40 to 52
Population: Randomized Population
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 879 | 872
g/dL | 1.52 (0.052) | 1.48 (0.053)
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Treatment comparison: Vadadustat minus Darbepoetin Alfa; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Least squares mean difference = 0.04, 95% CI 2-sided [-0.06 to 0.14], Standard Error of Mean 0.052

4. Secondary Outcome: Median Time to First MACE Plus Hospitalization for Heart Failure or Thromboembolic Event Excluding Vascular Access Thrombosis
Description: MACE was defined as all-cause mortality, non-fatal MI, or non-fatal stroke. Hospitalization for EAC adjudicated heart failure included presentation of participants to an acute care facility requiring an overnight hospitalization (change in calendar day) with an exacerbation of heart failure requiring treatment. EAC confirmed thromboembolic events for this secondary outcome measure included arterial thrombosis, deep vein thrombosis, and pulmonary embolism. PROTECT MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Results and statistical analysis from study AKB-6548-CI-0014 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0014 and AKB-6548-CI-0015 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to Week 208
Population: Safety Population (PRO2TECT). Only those participants with MACE plus hospitalization for heart failure or thromboembolic event excluding vascular access thrombosis were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 254 | 229
Weeks | 37.64 [17.14 to 74.14] | 41.43 [21.71 to 75.14]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0014 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.1743, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.966 to 1.382]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Time to first MACE plus hospitalization for heart failure or thromboembolic events excluding vascular access thrombosis for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 451 and 424 respectively; median time to first event (Q1, Q3) = 42.86 (19.71, 73.43) weeks versus 43.86 (21.36, 80.43) weeks, respectively; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.2305, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.972 to 1.267]

5. Secondary Outcome: Median Time to First Cardiovascular MACE
Description: MACE was defined as all-cause mortality, non-fatal MI, or non-fatal stroke. Cardiovascular MACE analysis differed from the primary MACE endpoint as it included only deaths adjudicated by the EAC as cardiovascular deaths (i.e, only EAC-confirmed cardiovascular deaths) in addition to first events of non-fatal MI or non-fatal stroke. PROTECT MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Results and statistical analysis from study AKB-6548-CI-0014 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0014 and AKB-6548-CI-0015 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to Week 208
Population: Safety Population (PRO2TECT). Only those participants with cardiovascular MACE events were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 109 | 95
Weeks | 45.86 [22.29 to 78.86] | 41.86 [20.29 to 90.00]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0014 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.3154, Gray's Test; Based on non-parametric analysis; Hazard Ratio (HR) = 1.19, 95% CI 2-sided [0.901 to 1.564]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Time to first cardiovascular MACE for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 198 and 178 respectively; median time to first event (Q1, Q3) = 45.57 (21.71, 73.29) weeks versus 47.36 (20.00, 88.43) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.2531, Gray's Test; Based on non-parametric analysis; Hazard Ratio (HR) = 1.16, 95% CI 2-sided [0.947 to 1.420]

6. Secondary Outcome: Median Time to First Cardiovascular Death
Description: Cardiovascular death included EAC adjudicated fatal MI, pump failure, sudden death, presumed sudden death, fatal stroke, fatal pulmonary embolism, cardiovascular procedure-related death, other cardiovascular death, and presumed cardiovascular death. PROTECT MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Results and statistical analysis from study AKB-6548-CI-0014 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0014 and AKB-6548-CI-0015 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to Week 208
Population: Safety Population (PRO2TECT). Only those participants with cardiovascular death were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 71 | 65
Weeks | 48.29 [28.86 to 83.14] | 41.86 [16.00 to 92.29]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0014 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.5991, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 1.13, 95% CI 2-sided [0.808 to 1.594]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Time to first cardiovascular death for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 127 and 131 respectively; median time to first event (Q1, Q3) = 48.29 (28.86, 76.14) weeks versus 48.43 (21.29, 92.29) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.8613, Gray's test; Based on non-parametric analysis; Hazard Ratio (HR) = 1.01, 95% CI 2-sided [0.792 to 1.293]

7. Secondary Outcome: Median Time to First All-cause Mortality
Description: Only events that were positively adjudicated and confirmed by the EAC were included in the MACE analyses. PROTECT MACE results and analysis, by design, was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Results and statistical analysis from study AKB-6548-CI-0014 has been reported in below table and under section "Statistical Analysis 1". Results and statistical analysis of the pooled data from studies AKB-6548-CI-0014 and AKB-6548-CI-0015 has been reported under section "Statistical Analysis 2" of this outcome measure.
Time Frame: Up to Week 208
Population: Safety Population (PRO2TECT). Only those participants with all-cause mortality were analyzed for this outcome measure.
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | Vadadustat | Darbepoetin Alfa
Number analyzed (Participants) | 180 | 168
Weeks | 46.57 [22.29 to 84.36] | 47.79 [27.36 to 88.79]
Statistical Analysis 1: Comparison: Vadadustat vs Darbepoetin Alfa; Statistical analysis from study AKB-6548-CI-0014 has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.4388, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.11, 95% CI 2-sided [0.902 to 1.375]
Statistical Analysis 2: Comparison: Vadadustat vs Darbepoetin Alfa; MACE analysis was performed on pooled data from studies AKB-6548-CI-0014 (NCT02648347) and AKB-6548-CI-0015 (NCT02680574). Time to first all-cause mortality for the Vadadustat and Darbepoetin alfa treatment groups was as follows: participants with events = 319 and 307 respectively; median time to first event (Q1, Q3) = 52.14 (28.71, 84.71) weeks versus 53.00 (30.71, 94.14) weeks, respectively. Statistical analysis from the pooled data has been reported in this section; Test type: Non-Inferiority — The prespecified non-inferiority margin was 1.25 (per FDA) and 1.3 (per EMA); p = 0.4577, Log Rank; Based on non-parametric analysis; Hazard Ratio (HR) = 1.09, 95% CI 2-sided [0.930 to 1.274]

8. Other Pre Specified Outcome: Exploratory - Proportion of Participants With Hb Values Within the Target Range During the Primary Evaluation Period (Weeks 24 to 36)
Time Frame: Weeks 24 to 36
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Exploratory - Proportion of Time With Hb Values Within the Target Range During the Primary Evaluation Period (Weeks 24 to 36)
Time Frame: Weeks 24 to 36
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Exploratory - Proportion of Time With Hb Values Within the Target Range During the Secondary Evaluation Period (Weeks 40 to 52)
Time Frame: Weeks 40 to 52
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Exploratory - Proportion of Participants With Hb Values Within the Target Range During the Secondary Evaluation Period (Weeks 40 to 52)
Time Frame: Weeks 40 to 52
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Exploratory - Proportion of Participants With an Hb Increase of >1.0 g/dL From Baseline Visit
Time Frame: Baseline; up to Week 52
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Exploratory - Time to Achieve Hb Increase of >1.0 g/dL From Baseline Visit
Time Frame: Baseline; up to Week 52
Reporting Status: Not Posted

14. Other Pre Specified Outcome: Exploratory - Mean Change in Hb Between Baseline (Mean Pretreatment Hb) and the Primary Evaluation Period (Mean Hb From Weeks 24 to 36) Stratified by Pre-baseline Erythropoiesis-stimulating Agent (ESA) Exposure
Time Frame: Baseline; Weeks 24 to 36
Reporting Status: Not Posted

15. Other Pre Specified Outcome: Exploratory - Mean Monthly Dose of Intravenous (IV) Elemental Iron Administered in Participants Who Have Received IV Iron
Time Frame: Up to Week 52
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Exploratory - Proportion of Participants Receiving IV Iron Therapy
Time Frame: Up to Week 52
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Exploratory - Proportion of Participants Receiving Red Blood Cells (RBCs) Transfusion(s)
Time Frame: Up to Week 52
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 208 weeks
Description: Treatment-emergent adverse events (TEAEs), defined as adverse events (AEs) that began (or pre-existing AEs that worsened) on or after the first dose through each participant's last participation date, were reported in study AKB-6548-CI-0014 (NCT02648347). Of the participants randomized, 1748 participants were included in the Safety population (878 and 870 participants in the Vadadustat and Darbepoetin alfa treatment groups, respectively). Three randomized participants did not receive treatment.
Arm/Group | Vadadustat | Darbepoetin Alfa
All-Cause Mortality (participants affected / at risk) | 180/878 | 168/870
Serious Adverse Events (participants affected / at risk) | 573/878 | 561/870
Other Adverse Events (participants affected / at risk) | 561/878 | 565/870
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vadadustat (N=878) | Darbepoetin Alfa (N=870)
End stage renal disease (Renal and urinary disorders) | 292 | 292
Pneumonia (Infections and infestations) | 60 | 49
Acute kidney injury (Renal and urinary disorders) | 42 | 40
Cardiac failure congestive (Cardiac disorders) | 40 | 39
Acute myocardial infarction (Cardiac disorders) | 32 | 27
Fluid overload (Metabolism and nutrition disorders) | 34 | 22
Sepsis (Infections and infestations) | 28 | 19
Hyperkalaemia (Metabolism and nutrition disorders) | 20 | 26
Cardiac failure acute (Cardiac disorders) | 21 | 24
Anaemia (Blood and lymphatic system disorders) | 18 | 24
Death (General disorders) | 23 | 19
Cardiac arrest (Cardiac disorders) | 23 | 16
Hypoglycaemia (Metabolism and nutrition disorders) | 18 | 20
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 15 | 18
Urinary tract infection (Infections and infestations) | 19 | 13
Cellulitis (Infections and infestations) | 16 | 13
Cardiac failure (Cardiac disorders) | 15 | 12
Coronary artery disease (Cardiac disorders) | 12 | 12
Chronic kidney disease (Renal and urinary disorders) | 15 | 9
Septic shock (Infections and infestations) | 12 | 11
Cardio-respiratory arrest (Cardiac disorders) | 9 | 12
Fall (Injury, poisoning and procedural complications) | 12 | 9
Cerebrovascular accident (Nervous system disorders) | 9 | 12
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 8 | 13
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 10 | 10
Diabetic nephropathy (Renal and urinary disorders) | 8 | 12
Hypertensive urgency (Vascular disorders) | 9 | 11
Atrial fibrillation (Cardiac disorders) | 11 | 8
Metabolic encephalopathy (Nervous system disorders) | 9 | 10
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 7 | 11
Acute left ventricular failure (Cardiac disorders) | 8 | 9
Peritonitis (Infections and infestations) | 9 | 8
Azotaemia (Renal and urinary disorders) | 8 | 9
Blood loss anaemia (Blood and lymphatic system disorders) | 12 | 4
Hypertension (Vascular disorders) | 6 | 10
Dehydration (Metabolism and nutrition disorders) | 4 | 11
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 9 | 6
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Gastroenteritis (Infections and infestations) | 9 | 5
Osteomyelitis (Infections and infestations) | 6 | 8
Urosepsis (Infections and infestations) | 7 | 7
Syncope (Nervous system disorders) | 7 | 7
Myocardial infarction (Cardiac disorders) | 5 | 8
Gangrene (Infections and infestations) | 7 | 6
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 8 | 5
Hypertensive emergency (Vascular disorders) | 4 | 9
Hypotension (Vascular disorders) | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 9 | 3
Hip fracture (Injury, poisoning and procedural complications) | 5 | 7
Angina unstable (Cardiac disorders) | 3 | 8
Transaminases increased (Investigations) | 7 | 4
Metabolic acidosis (Metabolism and nutrition disorders) | 6 | 5
Ischaemic stroke (Nervous system disorders) | 5 | 6
Uraemic encephalopathy (Nervous system disorders) | 7 | 4
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 5 | 6
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 6 | 5
Nephrogenic anaemia (Blood and lymphatic system disorders) | 5 | 5
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 6
Renal failure (Renal and urinary disorders) | 9 | 1
Diabetic foot (Skin and subcutaneous tissue disorders) | 5 | 5
Asthenia (General disorders) | 9 | 0
Non-cardiac chest pain (General disorders) | 6 | 3
Influenza (Infections and infestations) | 6 | 3
Hypovolaemia (Metabolism and nutrition disorders) | 7 | 2
Transient ischaemic attack (Nervous system disorders) | 6 | 3
Deep vein thrombosis (Vascular disorders) | 6 | 3
Cardiac failure chronic (Cardiac disorders) | 3 | 5
Cardiogenic shock (Cardiac disorders) | 6 | 2
Clostridium difficile colitis (Infections and infestations) | 7 | 1
Staphylococcal sepsis (Infections and infestations) | 5 | 3
Femur fracture (Injury, poisoning and procedural complications) | 2 | 6
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 | 4
Mental status changes (Psychiatric disorders) | 4 | 4
Hypertensive crisis (Vascular disorders) | 2 | 6
Peripheral vascular disorder (Vascular disorders) | 4 | 4
Angina pectoris (Cardiac disorders) | 5 | 2
Left ventricular failure (Cardiac disorders) | 1 | 6
Gastritis (Gastrointestinal disorders) | 3 | 4
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 3
Bronchitis (Infections and infestations) | 3 | 4
Pneumonia bacterial (Infections and infestations) | 2 | 5
Pyelonephritis (Infections and infestations) | 2 | 5
Pelvic fracture (Injury, poisoning and procedural complications) | 3 | 4
Alanine aminotransferase increased (Investigations) | 3 | 4
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Device related infection (Infections and infestations) | 5 | 1
Diverticulitis (Infections and infestations) | 1 | 5
Escherichia urinary tract infection (Infections and infestations) | 5 | 1
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 3 | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 5
Aspartate aminotransferase increased (Investigations) | 3 | 3
Gout (Metabolism and nutrition disorders) | 4 | 2
Hepatic encephalopathy (Nervous system disorders) | 3 | 3
Glomerulonephritis (Renal and urinary disorders) | 2 | 4
Aortic stenosis (Vascular disorders) | 0 | 6
Peripheral arterial occlusive disease (Vascular disorders) | 4 | 2
Peripheral ischaemia (Vascular disorders) | 3 | 3
Ascites (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 3 | 2
Generalised oedema (General disorders) | 4 | 1
Cholecystitis acute (Hepatobiliary disorders) | 4 | 1
Bacteraemia (Infections and infestations) | 3 | 2
Localised infection (Infections and infestations) | 4 | 1
Postoperative wound infection (Infections and infestations) | 2 | 3
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 2 | 3
Femoral neck fracture (Injury, poisoning and procedural complications) | 3 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 5 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 4
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 3 | 2
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 2
Plasma cell myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 4
Device occlusion (Product Issues) | 3 | 2
Haematuria (Renal and urinary disorders) | 3 | 2
Hypertensive nephropathy (Renal and urinary disorders) | 2 | 3
Renal tubular necrosis (Renal and urinary disorders) | 3 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 3
Atrial flutter (Cardiac disorders) | 2 | 2
Bradycardia (Cardiac disorders) | 1 | 3
Supraventricular tachycardia (Cardiac disorders) | 2 | 2
Abdominal pain (Gastrointestinal disorders) | 4 | 0
Constipation (Gastrointestinal disorders) | 1 | 3
Impaired gastric emptying (Gastrointestinal disorders) | 2 | 2
Intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Pancreatitis acute (Gastrointestinal disorders) | 3 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 2
Uraemic gastropathy (Gastrointestinal disorders) | 3 | 1
Multiple organ dysfunction syndrome (General disorders) | 3 | 1
Hepatic cirrhosis (Hepatobiliary disorders) | 2 | 2
Abscess limb (Infections and infestations) | 1 | 3
Arthritis bacterial (Infections and infestations) | 3 | 1
Cystitis (Infections and infestations) | 3 | 1
Diabetic foot infection (Infections and infestations) | 1 | 3
Pyelonephritis acute (Infections and infestations) | 1 | 3
Pyelonephritis chronic (Infections and infestations) | 1 | 3
Staphylococcal bacteraemia (Infections and infestations) | 1 | 3
Urinary tract infection bacterial (Infections and infestations) | 3 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 2
Humerus fracture (Injury, poisoning and procedural complications) | 2 | 2
Hepatic enzyme increased (Investigations) | 2 | 2
Hypervolaemia (Metabolism and nutrition disorders) | 3 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 3
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 2
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Brain injury (Nervous system disorders) | 1 | 3
Device dislocation (Product Issues) | 1 | 3
Hydronephrosis (Renal and urinary disorders) | 2 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 3
Orthostatic hypotension (Vascular disorders) | 2 | 2
Pancytopenia (Blood and lymphatic system disorders) | 1 | 2
Arrhythmia (Cardiac disorders) | 3 | 0
Atrioventricular block complete (Cardiac disorders) | 2 | 1
Atrioventricular block second degree (Cardiac disorders) | 2 | 1
Pericardial effusion (Cardiac disorders) | 0 | 3
Sinus node dysfunction (Cardiac disorders) | 2 | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 2 | 1
Gastric ulcer (Gastrointestinal disorders) | 2 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 2 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 2
Mallory-Weiss syndrome (Gastrointestinal disorders) | 2 | 1
Obstructive pancreatitis (Gastrointestinal disorders) | 3 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 2 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 2 | 1
Chest pain (General disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 1
Cholelithiasis (Hepatobiliary disorders) | 2 | 1
Clostridium difficile infection (Infections and infestations) | 1 | 2
Peritonitis bacterial (Infections and infestations) | 2 | 1
Pulmonary sepsis (Infections and infestations) | 3 | 0
Viral infection (Infections and infestations) | 1 | 2
Subdural haematoma (Injury, poisoning and procedural complications) | 2 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 2
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 | 3
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 2
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 3 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 0
Myositis (Musculoskeletal and connective tissue disorders) | 1 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 1
Cerebral infarction (Nervous system disorders) | 1 | 2
Dizziness (Nervous system disorders) | 2 | 1
Embolic stroke (Nervous system disorders) | 2 | 1
Encephalopathy (Nervous system disorders) | 1 | 2
Generalised tonic-clonic seizure (Nervous system disorders) | 1 | 2
Haemorrhage intracranial (Nervous system disorders) | 3 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 3
Seizure (Nervous system disorders) | 2 | 1
Glomerulonephritis chronic (Renal and urinary disorders) | 1 | 2
Nephropathy toxic (Renal and urinary disorders) | 2 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 0
Extremity necrosis (Vascular disorders) | 1 | 2
Peripheral artery thrombosis (Vascular disorders) | 1 | 2
Shock haemorrhagic (Vascular disorders) | 3 | 0
Steal syndrome (Vascular disorders) | 1 | 2
Coagulopathy (Blood and lymphatic system disorders) | 1 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 1
Aortic valve stenosis (Cardiac disorders) | 1 | 1
Arteriosclerosis coronary artery (Cardiac disorders) | 2 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 1
Cardiomyopathy (Cardiac disorders) | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 2
Sinus bradycardia (Cardiac disorders) | 1 | 1
Ventricular extrasystoles (Cardiac disorders) | 2 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 2 | 0
Hyperthyroidism (Endocrine disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 2 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 1
Vitreous haemorrhage (Eye disorders) | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 2
Diabetic gastroparesis (Gastrointestinal disorders) | 2 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 1
Enteritis (Gastrointestinal disorders) | 1 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Haematochezia (Gastrointestinal disorders) | 2 | 0
Hiatus hernia (Gastrointestinal disorders) | 0 | 2
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 2 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 1
Peptic ulcer haemorrhage (Gastrointestinal disorders) | 0 | 2
Catheter site haemorrhage (General disorders) | 1 | 1
Device related thrombosis (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 2
Peripheral swelling (General disorders) | 1 | 1
Sudden death (General disorders) | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 2 | 0
Abdominal abscess (Infections and infestations) | 0 | 2
Arteriovenous fistula site infection (Infections and infestations) | 1 | 1
Cellulitis gangrenous (Infections and infestations) | 0 | 2
Cystitis klebsiella (Infections and infestations) | 2 | 0
Device related sepsis (Infections and infestations) | 2 | 0
Endocarditis (Infections and infestations) | 1 | 1
Escherichia sepsis (Infections and infestations) | 0 | 2
Gas gangrene (Infections and infestations) | 2 | 0
Hepatitis C (Infections and infestations) | 1 | 1
Infected skin ulcer (Infections and infestations) | 1 | 1
Osteomyelitis acute (Infections and infestations) | 2 | 0
Pneumonia influenzal (Infections and infestations) | 0 | 2
Pneumonia staphylococcal (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Rhinovirus infection (Infections and infestations) | 1 | 1
Staphylococcal infection (Infections and infestations) | 2 | 0
Urinary tract infection staphylococcal (Infections and infestations) | 0 | 2
Wound infection staphylococcal (Infections and infestations) | 2 | 0
Wound sepsis (Infections and infestations) | 1 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 2
Head injury (Injury, poisoning and procedural complications) | 1 | 1
Procedural pneumothorax (Injury, poisoning and procedural complications) | 1 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 2
Troponin increased (Investigations) | 1 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 1
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 2
Carotid arteriosclerosis (Nervous system disorders) | 0 | 2
Carotid artery stenosis (Nervous system disorders) | 0 | 2
Cerebrovascular disorder (Nervous system disorders) | 2 | 0
Dysarthria (Nervous system disorders) | 1 | 1
Lacunar infarction (Nervous system disorders) | 1 | 1
Presyncope (Nervous system disorders) | 0 | 2
Tremor (Nervous system disorders) | 2 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 2
Nephrotic syndrome (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 1
Urinary retention (Renal and urinary disorders) | 1 | 1
Urinary tract obstruction (Renal and urinary disorders) | 0 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 1 | 1
Accelerated hypertension (Vascular disorders) | 2 | 0
Diabetic vascular disorder (Vascular disorders) | 0 | 2
Dry gangrene (Vascular disorders) | 1 | 1
Haematoma (Vascular disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 1
Haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 0
Immune thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Leukaemoid reaction (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 1 | 0
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 | 0
Adams-Stokes syndrome (Cardiac disorders) | 0 | 1
Atrial tachycardia (Cardiac disorders) | 0 | 1
Atrioventricular block (Cardiac disorders) | 0 | 1
Bundle branch block (Cardiac disorders) | 1 | 0
Cardiac tamponade (Cardiac disorders) | 1 | 0
Cardiac valve disease (Cardiac disorders) | 1 | 0
Cardiomegaly (Cardiac disorders) | 0 | 1
Cardiovascular insufficiency (Cardiac disorders) | 1 | 0
Chronic left ventricular failure (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Coronary artery thrombosis (Cardiac disorders) | 0 | 1
Diastolic dysfunction (Cardiac disorders) | 0 | 1
Hypertensive heart disease (Cardiac disorders) | 0 | 1
Ischaemic cardiomyopathy (Cardiac disorders) | 0 | 1
Left ventricular dysfunction (Cardiac disorders) | 1 | 0
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Pericardial haemorrhage (Cardiac disorders) | 0 | 1
Pericarditis uraemic (Cardiac disorders) | 1 | 0
Pulseless electrical activity (Cardiac disorders) | 1 | 0
Right ventricular dysfunction (Cardiac disorders) | 1 | 0
Stress cardiomyopathy (Cardiac disorders) | 1 | 0
Systolic dysfunction (Cardiac disorders) | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0
Arteriovenous malformation (Congenital, familial and genetic disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 | 0
Blindness (Eye disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1
Eye haemorrhage (Eye disorders) | 0 | 1
Macular degeneration (Eye disorders) | 1 | 0
Uveitis (Eye disorders) | 1 | 0
Vision blurred (Eye disorders) | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1
Cyclic vomiting syndrome (Gastrointestinal disorders) | 1 | 0
Dieulafoy's vascular malformation (Gastrointestinal disorders) | 0 | 1
Diverticular perforation (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal (Gastrointestinal disorders) | 0 | 1
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Erosive oesophagitis (Gastrointestinal disorders) | 0 | 1
Gastric antral vascular ectasia (Gastrointestinal disorders) | 1 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1
Haemorrhagic erosive gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 1 | 0
Intestinal infarction (Gastrointestinal disorders) | 0 | 1
Intestinal ischaemia (Gastrointestinal disorders) | 1 | 0
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intussusception (Gastrointestinal disorders) | 0 | 1
Irritable bowel syndrome (Gastrointestinal disorders) | 0 | 1
Large intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 1
Mesenteric artery thrombosis (Gastrointestinal disorders) | 0 | 1
Odynophagia (Gastrointestinal disorders) | 0 | 1
Oesophageal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Pancreatic necrosis (Gastrointestinal disorders) | 0 | 1
Reflux gastritis (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Accidental death (General disorders) | 0 | 1
Cardiac death (General disorders) | 0 | 1
Chest discomfort (General disorders) | 1 | 0
Complication of device insertion (General disorders) | 1 | 0
Fatigue (General disorders) | 1 | 0
Hypothermia (General disorders) | 1 | 0
Impaired healing (General disorders) | 0 | 1
Malaise (General disorders) | 1 | 0
Oedema (General disorders) | 0 | 1
Pyrexia (General disorders) | 1 | 0
Sudden cardiac death (General disorders) | 0 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis acute (Hepatobiliary disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Non-alcoholic steatohepatitis (Hepatobiliary disorders) | 1 | 0
Anti-neutrophil cytoplasmic antibody positive vasculitis (Immune system disorders) | 0 | 1
Renal transplant failure (Immune system disorders) | 1 | 0
Abdominal sepsis (Infections and infestations) | 0 | 1
Abdominal wall abscess (Infections and infestations) | 1 | 0
Abscess (Infections and infestations) | 1 | 0
Abscess neck (Infections and infestations) | 0 | 1
Acute hepatitis C (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Appendicitis perforated (Infections and infestations) | 0 | 1
Arteriovenous graft site infection (Infections and infestations) | 0 | 1
Arthritis infective (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis viral (Infections and infestations) | 0 | 1
Bronchopulmonary aspergillosis (Infections and infestations) | 0 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 0 | 1
Catheter bacteraemia (Infections and infestations) | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 0 | 1
Cholecystitis infective (Infections and infestations) | 0 | 1
Chronic hepatitis B (Infections and infestations) | 0 | 1
Chronic sinusitis (Infections and infestations) | 0 | 1
Diarrhoea infectious (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 0 | 1
Emphysematous cystitis (Infections and infestations) | 0 | 1
Encephalitis brain stem (Infections and infestations) | 0 | 1
Encephalitis viral (Infections and infestations) | 1 | 0
Endocarditis bacterial (Infections and infestations) | 0 | 1
Endocarditis staphylococcal (Infections and infestations) | 0 | 1
Endophthalmitis (Infections and infestations) | 1 | 0
Enterococcal bacteraemia (Infections and infestations) | 0 | 1
Escherichia bacteraemia (Infections and infestations) | 1 | 0
Escherichia pyelonephritis (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 1 | 0
Gastroenteritis clostridial (Infections and infestations) | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1
Groin abscess (Infections and infestations) | 1 | 0
H1N1 influenza (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Immune reconstitution inflammatory syndrome associated tuberculosis (Infections and infestations) | 1 | 0
Infected fistula (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 1
Mastoiditis (Infections and infestations) | 0 | 1
Medical device site joint infection (Infections and infestations) | 0 | 1
Metapneumovirus infection (Infections and infestations) | 0 | 1
Necrotising fasciitis (Infections and infestations) | 0 | 1
Necrotising soft tissue infection (Infections and infestations) | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1
Otitis media acute (Infections and infestations) | 0 | 1
Overgrowth bacterial (Infections and infestations) | 1 | 0
Parotitis (Infections and infestations) | 0 | 1
Pelvic inflammatory disease (Infections and infestations) | 1 | 0
Perineal abscess (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Pneumococcal sepsis (Infections and infestations) | 1 | 0
Pneumonia cryptococcal (Infections and infestations) | 0 | 1
Prostatic abscess (Infections and infestations) | 0 | 1
Pseudomonal bacteraemia (Infections and infestations) | 0 | 1
Salmonellosis (Infections and infestations) | 0 | 1
Scrotal abscess (Infections and infestations) | 0 | 1
Soft tissue infection (Infections and infestations) | 0 | 1
Staphylococcal abscess (Infections and infestations) | 1 | 0
Stoma site cellulitis (Infections and infestations) | 1 | 0
Streptococcal sepsis (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Urogenital infection bacterial (Infections and infestations) | 0 | 1
Viral sepsis (Infections and infestations) | 1 | 0
Wound abscess (Infections and infestations) | 0 | 1
Wound infection (Infections and infestations) | 0 | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1 | 0
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Facial bones fracture (Injury, poisoning and procedural complications) | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0
Fractured sacrum (Injury, poisoning and procedural complications) | 1 | 0
Iatrogenic injury (Injury, poisoning and procedural complications) | 0 | 1
Keratorhexis (Injury, poisoning and procedural complications) | 0 | 1
Lisfranc fracture (Injury, poisoning and procedural complications) | 1 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 0 | 1
Patella fracture (Injury, poisoning and procedural complications) | 0 | 1
Pelvic bone injury (Injury, poisoning and procedural complications) | 0 | 1
Peritoneal dialysis complication (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 1
Postpericardiotomy syndrome (Injury, poisoning and procedural complications) | 1 | 0
Procedural dizziness (Injury, poisoning and procedural complications) | 0 | 1
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Procedural nausea (Injury, poisoning and procedural complications) | 1 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 0
Skin injury (Injury, poisoning and procedural complications) | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Splenic rupture (Injury, poisoning and procedural complications) | 0 | 1
Subdural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1
Traumatic haemothorax (Injury, poisoning and procedural complications) | 0 | 1
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Urinary tract stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Vascular access malfunction (Injury, poisoning and procedural complications) | 1 | 0
Vascular access site pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Vascular injury (Injury, poisoning and procedural complications) | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1
Vulvovaginal injury (Injury, poisoning and procedural complications) | 0 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0
Anticoagulation drug level above therapeutic (Investigations) | 1 | 0
Arteriogram carotid abnormal (Investigations) | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood creatine increased (Investigations) | 1 | 0
Blood glucose decreased (Investigations) | 1 | 0
Blood pressure increased (Investigations) | 0 | 1
Glomerular filtration rate decreased (Investigations) | 0 | 1
Heart rate irregular (Investigations) | 1 | 0
Hepatic enzyme abnormal (Investigations) | 1 | 0
Liver function test abnormal (Investigations) | 1 | 0
Pulmonary arterial pressure increased (Investigations) | 0 | 1
Acidosis (Metabolism and nutrition disorders) | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemic hyperosmolar nonketotic syndrome (Metabolism and nutrition disorders) | 1 | 0
Hyperosmolar state (Metabolism and nutrition disorders) | 0 | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 1
Hypoosmolar state (Metabolism and nutrition disorders) | 0 | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 1
Vitamin B1 deficiency (Metabolism and nutrition disorders) | 1 | 0
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Neuropathic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Adrenal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Astrocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Astrocytoma, low grade (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cervix carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Colon neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Intraductal papillary mucinous neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung carcinoma cell type unspecified recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastatic bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Non-small cell lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal squamous cell carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Papillary renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Plasma cell myeloma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectosigmoid cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Squamous cell carcinoma of lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Altered state of consciousness (Nervous system disorders) | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0
Autonomic neuropathy (Nervous system disorders) | 0 | 1
Basal ganglia infarction (Nervous system disorders) | 1 | 0
Brain oedema (Nervous system disorders) | 1 | 0
Brain stem haemorrhage (Nervous system disorders) | 1 | 0
Brain stem stroke (Nervous system disorders) | 0 | 1
Cerebellar stroke (Nervous system disorders) | 0 | 1
Cerebral arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Cerebral small vessel ischaemic disease (Nervous system disorders) | 1 | 0
Coma (Nervous system disorders) | 1 | 0
Focal dyscognitive seizures (Nervous system disorders) | 1 | 0
Guillain-Barre syndrome (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Hypertensive encephalopathy (Nervous system disorders) | 1 | 0
Hypoglycaemic encephalopathy (Nervous system disorders) | 0 | 1
Hypoglycaemic seizure (Nervous system disorders) | 0 | 1
Hyponatraemic seizure (Nervous system disorders) | 1 | 0
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 0 | 1
Myelopathy (Nervous system disorders) | 0 | 1
Myoclonus (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 1 | 0
Toxic encephalopathy (Nervous system disorders) | 0 | 1
VIth nerve paralysis (Nervous system disorders) | 0 | 1
Vascular dementia (Nervous system disorders) | 1 | 0 (0)
Device adhesion issue (Product Issues) | 1 | 0
Device malfunction (Product Issues) | 1 | 0
Bipolar disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 0
Psychotic disorder (Psychiatric disorders) | 1 | 0
Bladder outlet obstruction (Renal and urinary disorders) | 1 | 0
Bladder perforation (Renal and urinary disorders) | 1 | 0
Glomerulonephritis rapidly progressive (Renal and urinary disorders) | 0 | 1
Hydroureter (Renal and urinary disorders) | 1 | 0
IgA nephropathy (Renal and urinary disorders) | 1 | 0
Lupus nephritis (Renal and urinary disorders) | 0 | 1
Nephritic syndrome (Renal and urinary disorders) | 0 | 1
Obstructive nephropathy (Renal and urinary disorders) | 0 | 1
Post infection glomerulonephritis (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1
Renal artery stenosis (Renal and urinary disorders) | 0 | 1
Renal mass (Renal and urinary disorders) | 1 | 0
Renal tubular acidosis (Renal and urinary disorders) | 0 | 1
Ureteric obstruction (Renal and urinary disorders) | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 1
Balanoposthitis (Reproductive system and breast disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 1 | 0
Haemorrhagic ovarian cyst (Reproductive system and breast disorders) | 1 | 0
Uterine prolapse (Reproductive system and breast disorders) | 1 | 0
Varicocele (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Laryngeal oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic wound (Skin and subcutaneous tissue disorders) | 0 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 1
Ingrowing nail (Skin and subcutaneous tissue disorders) | 0 | 1
Physical disability (Social circumstances) | 1 | 0
Arteriovenous fistula operation (Surgical and medical procedures) | 0 | 1
Aortic aneurysm (Vascular disorders) | 0 | 1
Aortic aneurysm rupture (Vascular disorders) | 1 | 0
Aortic rupture (Vascular disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Circulatory collapse (Vascular disorders) | 0 | 1
Essential hypertension (Vascular disorders) | 1 | 0
Haemorrhage (Vascular disorders) | 1 | 0
Iliac artery perforation (Vascular disorders) | 1 | 0
Internal haemorrhage (Vascular disorders) | 0 | 1
Malignant hypertension (Vascular disorders) | 1 | 0
Peripheral artery stenosis (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 1 | 0
Subclavian artery stenosis (Vascular disorders) | 0 | 1
Vasculitis (Vascular disorders) | 1 | 0
Venous perforation (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vadadustat (N=878) | Darbepoetin Alfa (N=870)
Hypertension (Vascular disorders) | 151 | 186
Hyperkalaemia (Metabolism and nutrition disorders) | 93 | 121
Diarrhoea (Gastrointestinal disorders) | 114 | 85
Oedema peripheral (General disorders) | 110 | 89
Urinary tract infection (Infections and infestations) | 98 | 94
Nausea (Gastrointestinal disorders) | 87 | 71
Fall (Injury, poisoning and procedural complications) | 74 | 80
Constipation (Gastrointestinal disorders) | 74 | 72
Hyperphosphataemia (Metabolism and nutrition disorders) | 64 | 63
Upper respiratory tract infection (Infections and infestations) | 50 | 70
Vomiting (Gastrointestinal disorders) | 60 | 52
Metabolic acidosis (Metabolism and nutrition disorders) | 63 | 48
Cough (Respiratory, thoracic and mediastinal disorders) | 47 | 58
Fluid overload (Metabolism and nutrition disorders) | 45 | 55
Back pain (Musculoskeletal and connective tissue disorders) | 55 | 45
Nasopharyngitis (Infections and infestations) | 50 | 48
Hypoglycaemia (Metabolism and nutrition disorders) | 46 | 52
Hypotension (Vascular disorders) | 49 | 49
Arthralgia (Musculoskeletal and connective tissue disorders) | 45 | 47
Headache (Nervous system disorders) | 46 | 42
Dizziness (Nervous system disorders) | 45 | 34
Bronchitis (Infections and infestations) | 28 | 46

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2019-02-26): https://cdn.clinicaltrials.gov/large-docs/47/NCT02648347/Prot_000.pdf
  • Statistical Analysis Plan (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/47/NCT02648347/SAP_001.pdf